CLINICAL TRIAL: NCT04940338
Title: The Effect of Topical Corticosteroids and Topical NSAIDs Perioperatively on IL6 Levels in Aqueous Humor and on Incidence of PCME in Patients With NPDR
Brief Title: PCME Prevention in Patients With NPDR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Principal Investigator, Andjela Jukic, MD, ophthalmologist, FEBO, Klinički Bolnički Centar Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR ZAG 02/21 AG 8.1-16/183-2
Record Dates: First submitted 2021-06-14; First posted 2021-06-25 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cystoid Macular Edema Following Cataract Surgery
Keywords: Pseudophakic cystoid macular edema (PCME); Interleukin-6 (IL6); Central foveal subfield thickness (CFT); Spectral domain Optical coherence tomography (SD-OCT)
MeSH Terms: interventions — Ophthalmic Solutions; bromfenac; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The drug pipettes will be covered with tape by hospital pharmacy and put into marked envelopes. The blinding will be uncovered after analyzing the data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bromfenac (Experimental): Group 1 will receive topical bromfenac (0.9 mg/mL) 2x daily, 7 days before the surgery
  Interventions: Drug: Bromfenac Ophthalmic 0.09% Ophthalmic Solution; Procedure: Phacoemulsification surgery (PHACO)
- Dexamethasone (Experimental): Group 2 will receive topical dexamethasone (1mg/mL) 2x daily before the surgery
  Interventions: Drug: Dexamethasone Ophthalmic; Procedure: Phacoemulsification surgery (PHACO)
- Placebo (Placebo Comparator): Group 3 will receive topical placebo (artificial tears substitute) 2x daily before the surgery
  Interventions: Drug: Placebo; Procedure: Phacoemulsification surgery (PHACO)

INTERVENTIONS:
Drug: Bromfenac Ophthalmic 0.09% Ophthalmic Solution — topical bromfenac (0.9 mg/mL) 2x daily 7 days before the surgery
  Other Names: Bromfenac
  Arms: Bromfenac
Drug: Dexamethasone Ophthalmic — topical dexamethasone (1 mg/mL) 2x daily 7 days before the surgery
  Other Names: Dexamethasone
  Arms: Dexamethasone
Drug: Placebo — topical placebo (artificial tears substitute) 2x daily before the surgery
  Arms: Placebo
Procedure: Phacoemulsification surgery (PHACO) — About 0.1-0.2 mL of aqueous humor will be collected at the beginning of the cataract surgery (PHACO) through paracentesis, aqueous will then be transported in dry ice with a dedicated box to the laboratory and stored at -80C until the analysis. IL6 concentration will be analyzed with Human IL6 Quantikine Elisa kit (R&D System).

SUMMARY:
Pseudophakic cystoid macular edema (PCME), or Irvine-Gass syndrome, is retinal thickening of the macula, which usually develops within 3 months after surgery, with a peak incidence between 4 and 6 weeks. Despite recent improvements in surgical techniques, PCME remains one of the most common causes of visual decline following an uneventful cataract surgery. Symptoms of PCME usually are blurred vision, metamorphopsia, loss of contrast sensitivity, and central scotomas. PCME usually responds well to medical therapy or may resolve spontaneously but carries a risk of permanent vision loss or loss of contrast sensitivity. There is wide discrepancy in opinions about the most effective antiinflammatory drops for the prevention of PCME. Patients with diabetes mellitus (DM) have attracted special interest because of higher incidence of cataract and increased risk for developing CME after cataract surgery. The optimum antiinflammatory prophylaxis for PCME in patients with nonproliferative diabetic retinopathy (NPDR) remains unknown.

Purpose of this study is to determine the efficacy of topical bromfenac and topical dexamethasone on intraocular concentration of interleukin-6 (IL6) and the incidence of pseudophakic cystoid macular edema (PCME) after cataract surgery in patients with nonproliferative diabetic retinopathy (NPDR).

DETAILED DESCRIPTION:
There is no standardized, widely-acceptable, evidence-based prophylaxis and treatment protocols to prevent macular edema after cataract surgery (PCME).

Current leading theory of pathogenesis of PCME (Irvine Gass) involves inflammation caused by surgical trauma which induces the release of inflammatory mediators like cytokines, prostaglandins and other vasopermeability factors, which disrupt the blood-retinal barrier and cause leakage from perifoveal retinal capillaries and accumulation of extracellular fluid in outer plexiform and inner nuclear layers of the retina. Diabetes is significant risk factor for developing PCME and grows proportionately with the severity of the diabetic retinopathy (DR). DR is common complication of diabetes mellitus (DM) and affects one in three persons with DM. Interleukin-6 (IL6) is associated with many intraocular inflammatory diseases such as diabetic retinopathy and macular edema acting as a pro-inflammatory cytokine. Levels of IL6 in aqueous humor are correlated with the severity of DR and the severity of DME. IL6 probably plays a crucial role in the development of inflammation after cataract surgery. Macular edema is usually monitored by spectral domain optical coherence tomography (SD-OCT) which is suitable for detecting subtle macular changes as well as follow up after treatment. OCT provides an objective measurement of macular thickness that correlates well with visual impairment and can be useful in standardizing definitions of PCME.

Prevention of PCME after cataract surgery in patients with NPDR include preoperative treatment with steroids, intravitreal injections of anti-vascular endothelial growth factors, laser treatment and topical nonsteroidal anti-inflammatory drugs (NSAIDs).

This randomized, double blinded, placebo-controlled trial will be conducted at Clinic of Ophthalmology, University Hospital Center Zagreb, Croatia. Ninety (90) eyes with mild to moderate NPDR (EDTRS classification) and cataract grade II nuclear/cortical or posterior subcapsular (Lens Opacities Classification System III) who will undergo phacoemulsification with intraocular lens implantation will be divided into three groups. Group 1 will receive topical bromfenac, group 2 will receive topical dexamethasone and group 3 will receive topical placebo, 7 days preoperatively and 3 weeks postoperatively. All patients will receive standard regimen of topical steroid-antibiotic drops postoperatively. Macular edema is defined as central foveal subfield thickness (CFT) increase of 40% from baseline. On the day of the surgery aqueous humor samples (0.1-0.2 mL) will be taken and IL6 concentration will be analyzed. Central foveal subfield thickness (CFT) will be measured with spectral domain optical coherence tomography (SD-OCT) and analyzed 7 days prior to surgery, on the day of the surgery and on 1, 7, 30 and 90 postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of mild to moderate nonproliferative diabetic retinopathy (EDTRS) and
* senile cataract grade II nuclear/cortical or posterior subcapsular (LOCS III)

Exclusion Criteria:

* anterior segment pathology (pseudoexfoliation syndrome, corneal opacities),
* posterior segment pathology (diabetic macular edema, previous diabetic macular edema treatment, previous retinal photocoagulation therapy, age related macular degeneration, retinal vascular diseases or history of uveitis)
* intraoperative complications (posterior capsular rupture, vitreus loss, intraocular lens not implanted in the capsular bag),
* postoperative complications (leaking incision, increased intraocular pressure, corneal edema or inflammation),
* therapy for glaucoma,
* patients on antihypertensive therapy, topical or systemic NSAIDs or steroids,
* previous steroid responders or hypersensitivity to the NSAID drug class,
* previous ocular trauma and intraocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 concentration | up to 12 weeks
  IL6 concentration in aqueous humor will be analyzed with Human IL6 Quantikine Elisa kit R&D System

SECONDARY OUTCOMES:
Central foveal subfield thickness (CFT) measured by optical coherence tomography (OCT) | 7 days before the surgery, on the day of the surgery, on 1, 7, 30 and 90 postoperative day
  Macular thickness will be reported according to the EDTRS thickness map. Central foveal subfield thickness (CFT) corresponds to the mean macular thickness in the central 1.0 mm area measured by optical coherence tomography (OCT).

CONTACTS AND LOCATIONS:
Overall Officials: Andjela Jukic, MD, FEBO, Principal Investigator — Klinički Bolnički Centar Zagreb; Miro Kalauz, MD, PHD, Study Director — Klinički Bolnički Centar Zagreb
Locations (1):
- KBCZagreb, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yonekawa Y, Kim IK. Pseudophakic cystoid macular edema. Curr Opin Ophthalmol. 2012 Jan;23(1):26-32. doi: 10.1097/ICU.0b013e32834cd5f8. PMID 22134362
- [Background] Russo A, Costagliola C, Delcassi L, Parmeggiani F, Romano MR, Dell'Omo R, Semeraro F. Topical nonsteroidal anti-inflammatory drugs for macular edema. Mediators Inflamm. 2013;2013:476525. doi: 10.1155/2013/476525. Epub 2013 Oct 21. PMID 24227908
- [Background] Han JV, Patel DV, Squirrell D, McGhee CN. Cystoid macular oedema following cataract surgery: A review. Clin Exp Ophthalmol. 2019 Apr;47(3):346-356. doi: 10.1111/ceo.13513. PMID 30953417
- [Background] Flach AJ. The incidence, pathogenesis and treatment of cystoid macular edema following cataract surgery. Trans Am Ophthalmol Soc. 1998;96:557-634. No abstract available. PMID 10360304
- [Background] Guo S, Patel S, Baumrind B, Johnson K, Levinsohn D, Marcus E, Tannen B, Roy M, Bhagat N, Zarbin M. Management of pseudophakic cystoid macular edema. Surv Ophthalmol. 2015 Mar-Apr;60(2):123-37. doi: 10.1016/j.survophthal.2014.08.005. Epub 2014 Sep 2. PMID 25438734
- [Background] Chu CJ, Johnston RL, Buscombe C, Sallam AB, Mohamed Q, Yang YC; United Kingdom Pseudophakic Macular Edema Study Group. Risk Factors and Incidence of Macular Edema after Cataract Surgery: A Database Study of 81984 Eyes. Ophthalmology. 2016 Feb;123(2):316-323. doi: 10.1016/j.ophtha.2015.10.001. Epub 2015 Dec 8. PMID 26681390
- [Background] Yau JW, Rogers SL, Kawasaki R, Lamoureux EL, Kowalski JW, Bek T, Chen SJ, Dekker JM, Fletcher A, Grauslund J, Haffner S, Hamman RF, Ikram MK, Kayama T, Klein BE, Klein R, Krishnaiah S, Mayurasakorn K, O'Hare JP, Orchard TJ, Porta M, Rema M, Roy MS, Sharma T, Shaw J, Taylor H, Tielsch JM, Varma R, Wang JJ, Wang N, West S, Xu L, Yasuda M, Zhang X, Mitchell P, Wong TY; Meta-Analysis for Eye Disease (META-EYE) Study Group. Global prevalence and major risk factors of diabetic retinopathy. Diabetes Care. 2012 Mar;35(3):556-64. doi: 10.2337/dc11-1909. Epub 2012 Feb 1. PMID 22301125
- [Background] Kim SJ, Schoenberger SD, Thorne JE, Ehlers JP, Yeh S, Bakri SJ. Topical Nonsteroidal Anti-inflammatory Drugs and Cataract Surgery: A Report by the American Academy of Ophthalmology. Ophthalmology. 2015 Nov;122(11):2159-68. doi: 10.1016/j.ophtha.2015.05.014. Epub 2015 Jun 26. PMID 26123091
- [Background] Jittpoonkuson T, Garcia PM, Rosen RB. Correlation between fluorescein angiography and spectral-domain optical coherence tomography in the diagnosis of cystoid macular edema. Br J Ophthalmol. 2010 Sep;94(9):1197-200. doi: 10.1136/bjo.2009.170589. Epub 2009 Dec 3. PMID 19965832
- [Background] Dong N, Xu B, Wang B, Chu L. Study of 27 aqueous humor cytokines in patients with type 2 diabetes with or without retinopathy. Mol Vis. 2013 Aug 4;19:1734-46. Print 2013. PMID 23922491
- [Background] Yao Y, Li R, Du J, Long L, Li X, Luo N. Interleukin-6 and Diabetic Retinopathy: A Systematic Review and Meta-Analysis. Curr Eye Res. 2019 May;44(5):564-574. doi: 10.1080/02713683.2019.1570274. Epub 2019 Feb 4. PMID 30644770
- [Background] Funatsu H, Yamashita H, Noma H, Mimura T, Yamashita T, Hori S. Increased levels of vascular endothelial growth factor and interleukin-6 in the aqueous humor of diabetics with macular edema. Am J Ophthalmol. 2002 Jan;133(1):70-7. doi: 10.1016/s0002-9394(01)01269-7. PMID 11755841
- [Background] Malecaze F, Chollet P, Cavrois E, Vita N, Arne JL, Ferrara P. Role of interleukin 6 in the inflammatory response after cataract surgery. An experimental and clinical study. Arch Ophthalmol. 1991 Dec;109(12):1681-3. doi: 10.1001/archopht.1991.01080120065027. PMID 1841575
- [Background] Badaro E, Novais E, Prodocimo LM, Sallum JM. Spectral-domain optical coherence tomography for macular edema. ScientificWorldJournal. 2014;2014:191847. doi: 10.1155/2014/191847. Epub 2014 May 14. PMID 24963500
- [Background] Eriksson U, Alm A, Bjarnhall G, Granstam E, Matsson AW. Macular edema and visual outcome following cataract surgery in patients with diabetic retinopathy and controls. Graefes Arch Clin Exp Ophthalmol. 2011 Mar;249(3):349-59. doi: 10.1007/s00417-010-1484-9. Epub 2010 Sep 9. PMID 20827486
- [Background] Wittpenn JR, Silverstein S, Heier J, Kenyon KR, Hunkeler JD, Earl M; Acular LS for Cystoid Macular Edema (ACME) Study Group. A randomized, masked comparison of topical ketorolac 0.4% plus steroid vs steroid alone in low-risk cataract surgery patients. Am J Ophthalmol. 2008 Oct;146(4):554-560. doi: 10.1016/j.ajo.2008.04.036. Epub 2008 Jul 2. PMID 18599019
- [Background] Kim SJ, Bressler NM. Optical coherence tomography and cataract surgery. Curr Opin Ophthalmol. 2009 Jan;20(1):46-51. doi: 10.1097/icu.0b013e3283199162. PMID 19093330
- [Background] Wielders LHP, Schouten JSAG, Winkens B, van den Biggelaar FJHM, Veldhuizen CA, Murta JCN, Goslings WRO, Kohnen T, Tassignon MJ, Joosse MV, Henry YP, Nagy ZZ, Rulo AHF, Findl O, Amon M, Nuijts RMMA; ESCRS PREMED study group. Randomized controlled European multicenter trial on the prevention of cystoid macular edema after cataract surgery in diabetics: ESCRS PREMED Study Report 2. J Cataract Refract Surg. 2018 Jul;44(7):836-847. doi: 10.1016/j.jcrs.2018.05.015. PMID 30055692
- [Background] Laursen SB, Erichsen JH, Holm LM, Kessel L. Prevention of macular edema in patients with diabetes after cataract surgery. J Cataract Refract Surg. 2019 Jun;45(6):854-869. doi: 10.1016/j.jcrs.2019.04.025. PMID 31146934
- [Background] Mamalis N. Prevention of cystoid macular edema after cataract surgery. J Cataract Refract Surg. 2018 Apr;44(4):419-420. doi: 10.1016/j.jcrs.2018.04.010. No abstract available. PMID 29778103
- [Background] Sarfraz MH, Haq RI, Mehboob MA. Effect of topical nepafenac in prevention of macular edema after cataract surgery in patients with non-proliferative diabetic retinopathy. Pak J Med Sci. 2017 Jan-Feb;33(1):210-214. doi: 10.12669/pjms.331.11644. PMID 28367202